CLINICAL TRIAL: NCT05033860
Title: The Influence of Education During Waiting Time of Vaccination on the Knowledge Towards COVID-19 Among Chinese Residents: A Randomized Controlled Trial
Brief Title: The Influence of Education During Waiting Time of Vaccination on the Knowledge Towards COVID-19 Among Chinese Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-R087
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Knowledge, Attitudes, Practice
MeSH Terms: conditions — COVID-19; Behavior | interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: 1. Intervention group: leaflets containing knowledge of COVID-19 and vaccination were distributed, and questionnaire surveys were conducted afterwards.
  2. Control group: questionnaire surveys were conducted without leaflets distribution.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Leaflets containing knowledge of COVID-19 and vaccination were distributed, and questionnaire surveys were conducted afterwards.
  Interventions: Other: Read leaflets containing knowledge of COVID-19 and vaccination.
- Control group (No Intervention): Questionnaire surveys were conducted without leaflets distribution.

INTERVENTIONS:
Other: Read leaflets containing knowledge of COVID-19 and vaccination. — Leaflets containing knowledge of COVID-19 and vaccination were distributed, and participants are asked to read the leaflets.
  Arms: Intervention group

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a respiratory disease caused by a novel coronavirus, which has developed the global pandemic situation. The promotion of vaccination is an effective strategy to control the epidemic. A total of 19,5738,000 doses of COVID-19 vaccines have been reported in China until August 24th, 2021. During widespread vaccination, the education in COVID-19 prevention and vaccination for residents are also crucial. To figure out the influence of education during waiting time of vaccination, we have designed a randomized controlled trial and planned to distribute leaflets and questionnaires to the residents of Xidian (a town in Ninghai, Zhejiang). This study is of great significance for the prevention of COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18;
2. Residents who are vaccinated with COVID-19 vaccines at Xidian Passenger Station from August 18th to September 20th, 2021;
3. Able to understand the content of leaflets and questionnaires, and willing to participate in the study.

Exclusion Criteria:

1. Residents who are unable to get vaccinated with COVID-19 vaccines;
2. Unable to understand the content of leaflets and questionnaires, or unwilling to participate in the study;
3. Unreturned or incomplete questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
Scores of the questionnaire | 5-20 minutes
  All the participants are asked to fulfill a questionnaire entitled "A survey on the public knowledge of COVID-19 and vaccination". The total score of questionnaire is calculated (full mark is 24). A higher score means a better knowledge of COVID-19 and vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No